CLINICAL TRIAL: NCT00764920
Title: Non-invasive Imaging Modalities for Assessment of Normal and Lesional Skin
Brief Title: Skin Imaging With Technologies in Development
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Kristen Kelly, Professor Departments of Dermatology and Surgery, University of California, Irvine
Other Study IDs: 20086307
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pigmented Skin Lesion of Uncertain Nature
Keywords: human skin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Skin Imaging: non-invasive imaging modalities for assessment of skin
  Interventions: Device: non-invasive imaging modalities for assessment of skin

INTERVENTIONS:
Device: non-invasive imaging modalities for assessment of skin — skin imaging

SUMMARY:
The purpose of this research is to develop non-invasive imaging modalities for assessment of skin. This is a pilot study which will use multiple imaging modalities to collect information on normal and lesional skin. The researchers understand that the purpose of this study is not to evaluate any particular treatment and an investigation of a new therapeutic intervention would require an additional protocol. Skin conditions to be studied include vascular lesions, pigmentary disorders, inflammatory conditions and neoplasms.

DETAILED DESCRIPTION:
Normal and lesional skin will be assessed by the following imaging modalities:

1. Laser Speckle Imaging can provide information about relative blood flow in a tissue. In skin it can be used to determine what areas have more blood flow and whether a particular intervention or treatment affects blood flow.
2. Optical Coherence Tomography and Optical Doppler Tomography can provide pictures of blood vessels in an area of the body and can also tell how fast blood is flowing in that area.
3. Photon Migration Spectroscopy can provide information about the amount of blood, oxygen, fat and water is in a tissue.
4. Multi-Spectral Imaging can provide a 3 dimensional image of structures within the skin.
5. Multiphoton Microscopy can provide images of structures of the skin.

ELIGIBILITY:
Inclusion Criteria:

* adult male or female 7 and older; able to carry out study instructions

Exclusion Criteria:

* Younger than 7 years old
* pregnant woman
* breast feeding

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be selected from University of California Irvine Medical Clinic
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2008-10; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Collect information on normal and lesional skin | up to 12 weeks
  Develop non-invasive imaging modalities for assessment of skin.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Kelly, MD, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute Medical Clinic, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No